CLINICAL TRIAL: NCT05339529
Title: Protective Effect of Thymosin Α1 Against Negative Immune Dysregulation and Organ Dysfunction After Acute Aortic Dissection Surgery (PANDA II)
Acronym: PANDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: Beijing Anzhen Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Qilu Hospital of Shandong University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Northern Jiangsu People's Hospital (Other); Guangdong Provincial People's Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Nanjing First Hospital, Nanjing Medical University (Other); Shanghai East Hospital,Tongji University School of Medicine (Unknown); The Seventh Affiliated Hospital of Xinjiang Medical University (Unknown); TEDA International Cardiovascular Hospital (Other); The First Affiliated Hospital of Bengbu Medical University (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PANDA II
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Acute Aortic Syndrome; Aortic Dissection Type a
MeSH Terms: conditions — Acute Aortic Syndrome | interventions — Thymalfasin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thymosin alpha 1 (Experimental): 1.6 mg q12h for 5 days
  Interventions: Drug: Thymosin Alpha1, 28A-Glycine-28B-L-Arginine-28C-L-Glutamic Acid-28D-L-Alanine-28E-L-Proline-28F-L-Alanine-28G-L-Asparagine-
- Blank control (Sham Comparator)
  Interventions: Drug: Blank control

INTERVENTIONS:
Drug: Thymosin Alpha1, 28A-Glycine-28B-L-Arginine-28C-L-Glutamic Acid-28D-L-Alanine-28E-L-Proline-28F-L-Alanine-28G-L-Asparagine- — Thymosin alpha 1, 1.6mg injection hypodermic (I.H), every 12 hours for 5 days at least during the ICU admission. The administration will be terminated any day during the treatment when the patient is deemed as qualified for ICU discharge or dead.
  Arms: Thymosin alpha 1
Drug: Blank control — Blank control
  Arms: Blank control

SUMMARY:
Systemic inflammatory response syndrome (SIRS) and multiple organ dysfunction syndrome (MODS) are the major causes of death in patients with acute aortic syndrome (AAS). Therefore, the prevention of SIRS and MODS is of great clinical value, and immunomodulatory therapy with thymosin alpha 1 may be beneficial. This study was designed to test the hypothesis that the administration of thymosin alpha 1 during the acute phase of AAS will result in a reduced incidence of SIRS and MODS.

ELIGIBILITY:
Inclusion Criteria:

* The patients are conformed to 2010 ACC/AHA guidelines for the diagnosis and treatment of thoracic aortic disease (TAD) within two weeks of onset;
* Patients with acute aortic syndrome confirmed clinically and radiologically and planning to undergo emergency surgery were enrolled.
* The patients' age between 18 ~90 years old.
* Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Patients allergic to Thymosin α1;
* Lactating women and pregnant women;
* Patients with mental diseases, drug and alcohol dependence;
* Refuse to participate in this study and refuse to sign the informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The highest Sequential Organ Failure Assessment (SOFA) score of 7 days after surgery | 7 days after surgery
  The occurrence of new-onset organ failure and new-onset persistent organ failure (Sequential Organ Failure Assessment (SOFA) score. New-onset is defined as events that occur after randomization and not present 24 hours before randomization.

SECONDARY OUTCOMES:
30-day mortality | 30 days after randomization
  Death from any cause of 30 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, Principal Investigator — Nanjing Medical University
Locations (15):
- China (15):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital Nanjing Medical University, Nanjing, Jiangsu
  - Subei People's Hospital of Jiangsu Province, Yangzhou, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Friendship Hospital of Yili Kazak Autonomous Prefecture, Kazak, Xinjiang
  - The Seventh Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Beijing Anzhen Hospital Capital Medical University, Beijing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Shanghai East Hospital Tongji University, Shanghai
  - TEDA International Cardiovascular Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu H, Qian SC, Zhang YY, Tang CB, Yue HH, Fan GL, Zhao X, Jiang YY, Huang FH, Zeng ZH, Wang W, Lu XR, Luo XK, Bai XF, Zheng XX, Xie P, Ma C, Zhao S, Zhang HJ; On the behalf of China Additive Anti-inflammatory Actions for Aortopathy and Arteriopathy (5A) and PANDA Trial Investigators. Effect of thymosin alpha1 on Immune response and organ function in acute aortic dissection surgery: PANDA II trial protocol. Future Cardiol. 2025 Jun;21(7):447-454. doi: 10.1080/14796678.2025.2505401. Epub 2025 May 14. PMID 40367062